CLINICAL TRIAL: NCT04121858
Title: Brain Safe: Consumer Intervention to Reduce Exposure to Drugs Linked to Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Richard Holden, Associate Professor, Indiana University School of Medicine Chief Healthcare Engineer, Center for Health Innovation and Implementation Science, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1811254189; R01AG056926 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Dementia
Keywords: anticholinergic; cognitive function; brain; aging
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Enroll 700 community-dwelling older adults who were prescribed one or more strong anticholinergics. Participants will be randomized to use the Brain Safe app or an attention control medication list app for 12 months, with monthly usage reminders.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator and outcome assessor will be masked to the App assignment (Brain Safe vs Attention Control Medication list App)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Safe App (Experimental): 1)Brain Safe App provides conversation starters for older adult patients on target anticholinergics. The conversation starters assist the patient to have discussions with their physicians regarding reduction in exposure to prescription anticholinergics. 2) Provides anticholinergic risk assessment.
  Interventions: Other: Brain Safe App
- Attention Control App (Sham Comparator): 1) Attention Control App provides a medication list for older patients to use but lacks the conversation starters for patient to use with there physicians aimed at reduction in exposure to prescription anticholinergics.2) No anticholinergic risk assessment.
  Interventions: Other: Attention Control App

INTERVENTIONS:
Other: Brain Safe App — The Brain Safe app includes the medication list, a personalized risk calculator, multimedia educational content, and a conversation starter/doctor's report.
  Arms: Brain Safe App
Other: Attention Control App — The attention control app, called Med Safe, includes only the medication list feature.
  Arms: Attention Control App

SUMMARY:
This study is an RCT to evaluate the effectiveness of Brain Safe on reducing anticholinergic exposure. Over 42 months, the trial will enroll 700 community-dwelling older adults who were prescribed one or more strong anticholinergics. Participants will be randomized to use the Brain Safe app or an attention control medication list app for 12 months, with monthly usage reminders.

DETAILED DESCRIPTION:
This study is a randomized clinical trial (RCT) of the efficacy of a direct-to-consumer intervention called Brain Safe to primarily reduce older adults' exposure to prescription anticholinergics and secondarily improve cognitive function and health-related quality of life. Over 42 months, the trial will enroll 700 community-dwelling older adults who were prescribed one or more strong anticholinergics. Participants will be randomized to use the Brain Safe app or an attention control medication list app for 12 months, with monthly usage reminders.

The primary objective is to test the effect of Brain Safe on anticholinergic exposure at 12 months. We hypothesize that anticholinergic exposure will be lower among those randomized to the Brain Safe intervention compared to those randomized to the attention control app at 12 months. Our primary, powered outcome is the total standard daily dose (TSDD) measure of anticholinergic exposure at 12 months, which is calculated over the preceding 6 months of prescription data. We will electronically capture prescription data monthly and compute TSDD at baseline, 6, and 12 months.

The secondary objective is to test the effect of Brain Safe on: (a) cognitive function and (b) health-related quality of life at 12 months. We hypothesize older adults randomized to Brain Safe will have higher (a) cognitive function, measured by using an objective, performance-based composite, and (b) health-related quality of life (HRQOL), compared to those randomized to the attention control app, at 12 months.

Exploratory objectives are to test the effect of Brain Safe on anticholinergic exposure, cognitive function, and HRQOL at 6 months. This aim will explore the presence of early effects of Brain Safe at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 1 primary care visit at Eskenazi Health or IU Health in past 12 months
* Age ≥ 60 years
* Written informed consent and HIPAA authorization for the release of personal health information.
* English-speaking
* At least one prescription for a strong anticholinergic medication with Anticholinergic Cognitive Burden (ACB) score 2 or 3 in prior 12 months, and currently using it
* Community-dwelling in Central Indiana
* Not cognitively impaired
* Not terminally ill
* Not sensory impaired (after correction)

Exclusion Criteria:

* Permanent resident of an extended care facility (nursing home); independent or assisted senior care living is allowed if managing own medications.
* Diagnosis of Alzheimer's disease or related dementia (ADRD), determined by International Classification of Diseases (ICD)-9/ICD-10 codes or current use of a medication for ADRD
* Diagnosis of schizophrenia, bipolar disorder, or schizoaffective disorder defined by ICD-9/ICD-10 codes
* Involvement in another clinical trial that would prevent or interfere with study objectives
* Sensory or other impairment prohibiting the use of a mobile touchscreen device or other study activity (after correction)
* Not currently using anticholinergic medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Total standardized daily dose (TSDD) - from medical records | 12 months
  Total standardized daily dose (TSDD), the cumulative anticholinergic burden computed from medical record medication data over the prior 6 months
Total standardized daily dose (TSDD) - self-report medication inventory | 12 months
  Total standardized daily dose (TSDD), the cumulative anticholinergic burden computed from self-reported medication inventory data in the Brain Safe or attention control app

SECONDARY OUTCOMES:
Choice reaction time (CRT) | 12 months
  Computer-based assessment of choice reaction time (CRT), used with simple reaction time (SRT) to assess executive function
Simple Reaction Time (SRT) | 12 months
  Computer-based test, used with Choice Reaction Time (CRT) test to compute a score, to assess executive function
Digit-Symbol Substitution Test (DSST) | 12 months
  Paper-based digit-symbol substitution test, from WAIS-IV ( Wechsler Adult Intelligence Scale-IV) Coding, used to assess processing speed
Hopkins Verbal Learning Test (HVLT) | 12 months
  Paper-based list learning and recall test, used to assess memory.
Trail Making Test (TMT) Parts A and B | 12 months
  Paper-based test, used to assess executive function
Health Utilities Index (HUI) Mark 3 | 12 months
  Self-reported measure of health-related quality of life, producing a single score on a standardized utility values range from -0.36 for the HUI-3, respectively, to 1.00 with higher scores indicating better outcome

OTHER OUTCOMES:
Medication perceptions | 12 months
  9-item standardized survey of medication perceptions; developed in-house based on combination of Health Belief Model questionnaires and revised Patients' Attitudes Towards Deprescribing Questionnaire; responses on 5-point agreement scale from strongly agree to strongly disagree, items analyzed separately and as subscale averages (range 1-5, higher indicating more disagreement/less agreement)
Self-reported deprescribing behavior | 12 months
  4-item standardized survey of self-reported deprescribing behaviors, developed in-house, responses on 5-point agreement scale from strongly agree to strongly disagree, items analyzed separately (range 1-5, higher indicating more disagreement/less agreement)
System Usability Scale | 12 months
  10-item standardized survey of user-reported technology usability, based on revised System Usability Scale, with scale score computed ranging from 0-100, with 100 indicating highest possible perceived usability
Satisfaction with technology: 3-item standardized survey | 12 months
  3-item standardized survey of user-reported satisfaction with technology, based on satisfaction items from Technology Acceptance Model questionnaires, responses on 5-point agreement scale from strongly agree to strongly disagree, items analyzed separately and as scale average (range 1-5, higher indicating more disagreement/less agreement)
Technology use | 12 months
  Usage logs of technology use over time

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Holden, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - IU Health, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Derived] Abebe E, Campbell NL, Clark DO, Tu W, Hill JR, Harrington AB, O'Neal G, Trowbridge KS, Vallejo C, Yang Z, Bo N, Knight A, Alamer KA, Carter A, Valenzuela R, Adeoye P, Boustani MA, Holden RJ. Reducing anticholinergic medication exposure among older adults using consumer technology: Protocol for a randomized clinical trial. Res Social Adm Pharm. 2021 May;17(5):986-992. doi: 10.1016/j.sapharm.2020.10.010. Epub 2020 Oct 22. PMID 33773639
- [Derived] Hill JR, Harrington AB, Adeoye P, Campbell NL, Holden RJ. Going Remote-Demonstration and Evaluation of Remote Technology Delivery and Usability Assessment With Older Adults: Survey Study. JMIR Mhealth Uhealth. 2021 Mar 4;9(3):e26702. doi: 10.2196/26702. PMID 33606655

DOCUMENTS (1):
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04121858/ICF_000.pdf